CLINICAL TRIAL: NCT04654299
Title: Prospective Study Correlating External Biliary Stenting and Pancreatic Fistula Following Pancreaticoduodenectomy
Brief Title: Biliary Externalization After Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Gerardo Blanco-Fernández, Chief of Department, Universidad de Extremadura
Other Study IDs: 20201129
Record Dates: First submitted 2020-11-29; First posted 2020-12-04 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Postoperative Complications
Keywords: Pancreaticoduodenectomy; Pancreatic postoperative fistula
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- standard PD (ST-PD): Pancreacoduodenectomy with pancreatic-enteric reconstruction and standard hepaticojejunostomy
- PD with external biliary stent(PD-BS): Pancreacoduodenectomy with pancreatic-enteric reconstruction and hepaticojejunostomy with external biliary stent for externalization of bile fluid
  Interventions: Procedure: External biliary stent

INTERVENTIONS:
Procedure: External biliary stent — The biliary stent consisted of a multi-perforated, natural rubber tube, measuring 3.5 mm in diameter, that we placed transanastomotically, with exteriorization sited at 20 cm utilizing the Witzel jejunostomy approach
  Groups: PD with external biliary stent(PD-BS)

SUMMARY:
Postoperative pancreatic fistula(POPF) is the most common complication of pancreaticoduodenectomy (PD). Sometimes POPF is associated with biliary fistula(BF), or "mixed" fistula. The purpose of this study is to assess whether the severity of the fistulae, when present, is decreased with an external biliary stent in place.

DETAILED DESCRIPTION:
n this single-center study we analyze patients who underwent elective PD from January_2014 to December_2017. Patients are divided into two groups: standard PD (ST-PD)vs PD with external biliary stent(PD-BS). Demographic, preoperative, intraoperative, and postoperative variables will be analyze, including complications according to the Clavien-Dindo classification, and those specific to pancreatic surgeries, and mortality rates within 90 days of operation.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Patient age > 18 years old;
* Elective pancreaticoduodenectomy performed for primary pancreatic disease.

Exclusion Criteria:

* Pancreaticoduodenectomy with multivisceral resection (organ other than duodenum, pancreas, gallbladder, and bile duct);
* Patients with peritoneal or liver metastases found during surgery.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergo elective pancreaticoduodenectomy
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 90 days
  Any postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Blanco-Fernández, MD, PhD, Study Director — Universidad de Extremadura

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blanco-Fernandez G, Jaen-Torrejimeno I, De-Armas-Conde N, Rojas-Holguin A, Naharro JS, Castillo-Tunon JM, Lopez-Guerra D. Prospective Study Correlating External Biliary Stenting and Pancreatic Fistula Following Pancreaticoduodenectomy. J Gastrointest Surg. 2021 Nov;25(11):2881-2888. doi: 10.1007/s11605-021-04983-6. Epub 2021 Mar 25. PMID 33768426